CLINICAL TRIAL: NCT04165889
Title: Evaluation of the Establishment of a Hospital Medication Report for Pharmacists and General Practitioners
Brief Title: Hospital Medication Report
Acronym: EvalMedReport
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0434
Record Dates: First submitted 2019-11-13; First posted 2019-11-18 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Drug Related Problem
Keywords: hospitalized in internal medicine unit; adult patient; Medication Error; Clinical Pharmacist

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Drug Related Problem (DRP) is defined as an event that may potentially affect the health outcomes in the patients. DRPs can occur at all stages of the medication usage process starting from prescribing (included medication error and inappropriate prescription) to dispensing stage. Lack of follow-ups and reassessment of therapeutic outcomes may also contribute to DRPs. Pharmaceutical care is a co-operative activity in concert with other health care professionals and offered directly to the patient for improved quality use of medicines. Pharmaceutical care identifies and resolves actual or potential DRPs.

In our clinical practice, during the patient admission in internal medicine unit, a medication reconciliation process was conducted according to a validated protocol. The first step consists of getting the Best Possible Medication History (BPMH), defined as the most comprehensive list of all medications taken by the patient. The second step consists of comparing the BPMH with admission prescription made by the physician in charge. During pharmacist interview, pharmacist discussed about medication adherence and knowledge. The third step consists of characterizing, solving and documenting DRPs.

During the patient's hospitalization, the pharmacist participates at the medication prescription revision. At the discharge of hospitalization, a pharmaceutical standardised interview is carried out during which the pharmacist explains the modifications of treatments to the patient. During this interview, the hospital pharmacist updates the latest treatment changes. For patient with more than 65 years old and long-term affection (or patient with more than 75 years old with or without long-term affection) and 5 medications, the hospital pharmacist write a medication discharge report (MDR) to patient, community pharmacist and general practitioner.

For each medication, the investigators collected its name, dosage, dosage forms and frequency of administration. For each DRP, the investigators collected the type of DRP and the drug classes (according to anatomical therapeutic chemical classification system).

For each MDR, the investigators collected number of medication, number and type of DRP including inappropriate prescription.

ELIGIBILITY:
Inclusion criteria:

- Patients aged above 18 years old, admitted to the medicine unit during the study period and hospitalized for at least 24 hours

Exclusion criteria:

- NA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population was composed of patient hospitalized in Montpellier University hospital.
Sampling Method: Non-Probability Sample
Enrollment: 280 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
number of patients with MDR | 1 day
  number of patients with MDR

SECONDARY OUTCOMES:
number of patients with MDR and DRP | 1 day
  number of patients with MDR and DRP

CONTACTS AND LOCATIONS:
Overall Officials: Cyril BREUKER, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC